CLINICAL TRIAL: NCT03386461
Title: Effect of Exercise Training and Omega-3 Fatty Acids on Metabolic Health and Dysfunction of Adipose Tissue in Elderly
Brief Title: Effect of Exercise and Omega-3 on Metabolic Health in Elderly
Acronym: EXODYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Michaela Siklova, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AZV 16-29182A
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Metabolism Disorder; Adiposity; Inflammatory Response
Keywords: elderly; exercise training; adipose tissue; omega-3 polyunsaturated fatty acids; inflammation; diferentiation of preadipocytes
MeSH Terms: conditions — Metabolic Diseases; Obesity; Inflammation | interventions — Exercise; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: The exercise training intervention with or without omega-3 supplementation (Calanus oil) will be prescribed to non-trained sedentary elderly women
Who Masked: Participant, Care Provider
Masking Description: Two types of pills (calanus or placebo) will be prescribed to subjects, investigator will randomly assign the subjects to the arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + Omega 3 supplementation (Experimental): Subjects will be enrolled in physical activity program that consists of combined aerobic and resistive training 3 times a week for 4 months. Training will be supervised by physiotherapists experienced in exercise training of elderly (Senior Fitness, and Faculty of Physical Education and Sport). Subjects will take 5 capsules od Calanus oil (containing approx. 250 mg EPA and DHA per day).
  Interventions: Behavioral: Exercise training; Dietary Supplement: omega 3 supplementation
- Exercise + placebo (Placebo Comparator): Subjects will be enrolled in physical activity program that consists of combined aerobic and resistive training 3 times a week for 4 months. Training will be supervised by physiotherapists experienced in exercise training of elderly. Subjects will take 5 capsules od placebo per day (provided by Calanus oil company, containing sunflower oil).
  Interventions: Behavioral: Exercise training; Dietary Supplement: placebo

INTERVENTIONS:
Behavioral: Exercise training — Combined aerobic and resistive training 3 times a week for 4 months. The strength training will be performed at moderate intensity (i.e., 50-60% of RM), and moderate volume (i.e., 2 to 3 sets per exercise). Endurance training will be performed at moderate- to high-intensity (i.e., 60-85% of VO2max) in the form of continuous and interval training (for high intensities), respectively. The training intensity will be prescribed individually on the basis of the initial exercise testing. Subjects will be thoroughly instructed on effective home-based exercise and advised to exercise in total 5 days a week.
Dietary Supplement: omega 3 supplementation — Capsules with high content of omega 3 fatty acids (Calanus oil) will be taken every day with lunch meal. The content of omega-3 fatty acids (EPA, DHA) per day should reach 250 mg.
  Other Names: Calanus oil
  Arms: Exercise + Omega 3 supplementation
Dietary Supplement: placebo — Capsules with content of omega 6 fatty acids (sunflower oil) will be taken every day with lunch meal.
  Other Names: sunflower oil
  Arms: Exercise + placebo

SUMMARY:
The aim of this project is to investigate in elderly women, the effect of combined aerobic and resistive training and concomitant supplementation with omega-3 fatty acids on adipogenesis, metabolic functions and pro-inflammatory status of adipose tissue and on systemic metabolic profile.

DETAILED DESCRIPTION:
Aging is associated with development of disturbances of lipid and carbohydrate metabolism and with systemic pro-inflammatory state similarly to the alterations observed in obese individuals. Metabolic and immune dysfunction of adipose tissue has been suggested as an important contributing trigger to this condition. EXODYA project is a clinical study in elderly individuals that aims to establish benefits of lifestyle intervention and nutritional supplementation -either alone or in combination- for the amelioration of systemic and adipose tissue metabolic and immune disturbances. Effects of 4 months´ intervention with combined aerobic plus resistive exercise training and supplementation with omega-3 polyunsaturated fatty acids on systemic metabolic profile and molecular characteristics of adipose tissue will be investigated in elderly women. Thus, a proof-of-concept will be provided for novel recommendations and guidelines for lifestyle interventions in elderly population

ELIGIBILITY:
Inclusion Criteria:

* elderly women: age 60-80
* non-trained (without regular physical activity)
* BMI in the range of 25-30 kg/m2

Exclusion Criteria:

* diagnosed cancer, diabetes, liver and renal diseases, untreated hyper- or hypo-thyroidism, long term use of anti-inflammatory medication (anti-rheumatics and analgesics affecting cyclooxygenases (100 mg of anopyrin daily is acceptable), steroids and/or Omega-3 dietary supplements

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in adipose tissue inflammation | through study completion, an average of 1 year
  analysis of distribution of immune cells (flow cytometry analysis)
Change in adipose tissue inflammatory signalling | through study completion, an average of 1 year
  analysis of pro-resolving mediators (UPLC-MS/MS methodology)

SECONDARY OUTCOMES:
Change in insulin sensitivity | through study completion, an average of 1 year
  Hyperinsulinemic izoglycemic clamp (GDR-glucose disposal rate)
Change in physical performance | through study completion, an average of 1 year
  Maximum graded exercise test on bicycle ergometer (Vo2max)
Change in gene expression in adipose tissue | through study completion, an average of 1 year
  mRNA expression of metabolic and inflammatory genes in adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Siklova, PhD, Principal Investigator — Third faculty of medicine, Charles University in Prague
Locations (1):
- Third Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cizkova T, Stepan M, Dadova K, Ondrujova B, Sontakova L, Krauzova E, Matous M, Koc M, Gojda J, Kracmerova J, Stich V, Rossmeislova L, Siklova M. Exercise Training Reduces Inflammation of Adipose Tissue in the Elderly: Cross-Sectional and Randomized Interventional Trial. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa630. doi: 10.1210/clinem/dgaa630. PMID 32902644
- [Derived] Brezinova M, Cajka T, Oseeva M, Stepan M, Dadova K, Rossmeislova L, Matous M, Siklova M, Rossmeisl M, Kuda O. Exercise training induces insulin-sensitizing PAHSAs in adipose tissue of elderly women. Biochim Biophys Acta Mol Cell Biol Lipids. 2020 Feb;1865(2):158576. doi: 10.1016/j.bbalip.2019.158576. Epub 2019 Nov 16. PMID 31740387